CLINICAL TRIAL: NCT01675362
Title: A Randomized Controlled Trial for Evaluating Protective Effects of Antioxidants (Selenium and Vitamins A, C and E), Calcium Channel Blocker (Verapamil) and Angiotensin Receptor Blocker (Losartan) Against Extracorporeal Shockwaves Lithotripsy Induced Renal Injury
Brief Title: Are There Protective Effects of Antioxidants, Calcium Channel Blocker and Angiotensin Receptor Blocker Against Extracorporeal Shockwaves Lithotripsy Induced Renal Injury?
Acronym: SWL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed R. EL-Nahas, Assistant Professor of Urology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4228
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Kidney Calculi
Keywords: Extracorporeal shockwave lithotripsy (ESWL); Kidney calculi; Renal protection; Antioxidants; Calcium channel blockers; Angiotensin receptor blockers
MeSH Terms: conditions — Kidney Calculi | interventions — Calcium Channel Blockers; Verapamil; Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control group (Placebo Comparator): They will receive placebo
  Interventions: Drug: Placebo
- Antioxidant group (Active Comparator): They will be receive vitamins A, C, E and selenium (Selenium ACE) Dosage: Two tablets before ESWL Then 2 tablets every 8 hours after ESWL for one week
  Interventions: Drug: Antioxidant group
- Calcium channel Blockers (Active Comparator): They will receive Verapamil (Isoptin 80 mg) Dosage: One tablet 2 hours before ESWL Then one tablet every 12 hours after ESWL for one week
  Interventions: Drug: Calcium Channel Blockers
- Angiotensin receptor blocker group (Active Comparator): They will receive Losartan (Cozaar 50 mg) Dosage: One tablet 2 hours before ESWL Then one tablet every day after ESWL for one week
  Interventions: Drug: Angiotensin receptor blocker group

INTERVENTIONS:
Drug: Antioxidant group — They will be receive vitamins A, C, E and selenium (Selenium ACE) Dosage: Two tablets before ESWL Then 2 tablets every 8 hours after ESWL for one week
  Other Names: Selenium ACE
  Arms: Antioxidant group
Drug: Calcium Channel Blockers — They will receive Verapamil (Isoptin 80 mg) Dosage: One tablet 2 hours before ESWL Then one tablet every 12 hours after ESWL for one week
  Other Names: Verapamil
  Arms: Calcium channel Blockers
Drug: Angiotensin receptor blocker group — They will receive Losartan (Cozaar 50 mg) Dosage: One tablet 2 hours before ESWL Then one tablet every day after ESWL for one week
  Other Names: Losartan
  Arms: Angiotensin receptor blocker group
Drug: Placebo — They will receive placebo
  Arms: Control group

SUMMARY:
This study will be conducted to evaluate the protective effects and mechanisms of antioxidants (vitamins A, C, E and Selenium), calcium channel blocker (Verapamil) and angiotensin receptor blocker (Lozartan) against shock wave induced renal injuries.

DETAILED DESCRIPTION:
The protective effect will be evaluated via estimation of the changes in renal tubular enzyme (NGAL) and detection of albumen levels in urine. The mechanisms of protection will be investigated by estimation of renal perfusion and functional changes using dynamic MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Well functioning kidney (serum creatinine <1.2 mg/dl).
2. Solitary renal stone.
3. Size: 25 mm or less in the largest diameter.

Exclusion Criteria:

1. Contraindications to ESWL
2. Previous surgical treatment of renal stones.
3. Congenital renal anomalies.
4. Pediatric patients (age <18 years).
5. Patients with Diabetes or hypertension

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Renal damage | two hours and one week after Extracorporeal shock wave lithotripsy (ESWL)
  The protective effect will be evaluated via estimation of the changes in renal tubular enzyme (NGAL) and detection of albumen levels in urine.

SECONDARY OUTCOMES:
The mechanisms of renal protection | Before ESWL, 2 hours and 1 week after ESWL
  The mechanisms of protection will be investigated by estimation of renal perfusion and functional changes using dynamic MRI

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed R. EL-Nahas, MD, Principal Investigator — Mansoura University
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Egypt